CLINICAL TRIAL: NCT01194596
Title: Effectiveness of Smoking Cessation Advice Combined With a Detailed Discussion of the Spirometric Results With the Primary Care Practitioner on the Smoking Habit in Adult Smokers (ESPITAP)
Brief Title: Effectiveness of Smoking Cessation Advice Combined With Spirometric Results in Adult Smokers (ESPITAP)
Acronym: ESPITAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Catalan Institute of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4R07/040; Jordi Gol i Gurina Foundation (Other: 4R07/040)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Smoking Cessation
Keywords: smoking cessation advice; spirometry; primary health care
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spirometry and lifestyle counseling (Experimental): Intervention group: will be given a brief but structured smoking cessation advice (according to the standards of the Tobacco Study Group of the Catalan Society of Family Medicine) together with a detailed and structured discussion of the spirometric results.
  Interventions: Behavioral: Smoking cessation advice; Behavioral: Spirometry and smoking cessation advice
- Lifestyle counseling (No Intervention): No intervention group: will be given a brief but structured smoking cessation advice (according to the standards of the Tobacco Study Group of the Catalan Society of Family Medicine).

INTERVENTIONS:
Behavioral: Smoking cessation advice — Brief but structured smoking cessation advice (according to the standards of the Tobacco Study Group of the Catalan Society of Family Medicine), will be given in both arms.
  Other Names: Usual care; Intervention arm; No Intervention arm
  Arms: Spirometry and lifestyle counseling
Behavioral: Spirometry and smoking cessation advice — Intervention group: will be given a brief but structured smoking cessation advice (according to the standards of the Tobacco Study Group of the Catalan Society of Family Medicine) together with a detailed and structured discussion of the spirometric results.
  Other Names: Intervention arm
  Arms: Spirometry and lifestyle counseling

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the spirometric results information advice about the smoking habit the investigators designed an intervention trial in primary care.

Hypothesis: In adult smokers, smoking cessation advice combined with a discussion of the spirometric tests on the part of the practitioner achieves a higher rate of tobacco reduction and abandonment than just smoking cessation advice.

Expected results: In adult smokers, a detailed discussion of the results yielded by spirometry tests together with brief smoking cessation advice on the part of the primary care practitioner can facilitate tobacco reduction and abandonment.

DETAILED DESCRIPTION:
Main objective: To evaluate the effectiveness of smoking cessation advice combined with a detailed discussion of the spirometric results with the primary care practitioner on the smoking habit in adult smokers.

Methodology:

Design: Intervention study using a randomised control group. Setting: 12 primary care centres of two health areas. Participants: 600 smokers, aged 35 to 70 years, seeking medical advice from their primary care practitioner (GP) for any given reason (selection visit), excluding those patients with Chronic Obstructive Pulmonary Disease (COPD).

Measurements and interventions: In the selection visit, all participants will be required to undergo a series of tests that will include spirometry, tobacco dependence test, a test to measure the motivation to stop smoking and a structured questionnaire on sociodemographic data, smoking habit, respiratory symptomatology, etc. Based on the spirometric results, patients presenting airflow limitation will be excluded.

Randomisation will be performed using a computer programme. Randomisation will be carried out by the Coordinating Centre.

All other patients will be scheduled for another visit with their primary care practitioner one month later. In this visit (visit 1) and depending on the randomisation into 2 groups, one group will be given brief but structured smoking cessation advice together with a detailed and structured discussion of the spirometric results while the second group will also be given the same brief smoking cessation advice but without discussing the spirometric results. Both groups will be scheduled for a visit at 6 months (visit 2), and at 1 year (visit 3). During visit 2, the patient will be asked about his or her smoking habit. One month before visit 3, patients will be required to undergo again the series of tests performed prior to visit 1. In visit 3, all those patients who claim to have stopped smoking will be required to take a carbon monoxide test.

ELIGIBILITY:
Inclusion Criteria:

* Adult smoker subjects aged between 35 and 70 years

Exclusion Criteria:

* Previous antecedents of any respiratory disease
* Suffering of any chronic or terminal disorder
* Counterindication to undertake spirometry or that may hinder the performance of the spirometry test

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
smoking abstinence: self reported abstinence (12 or more months) | 12 months
  smoking abstinence confirmed by an expired air carbon monoxide

SECONDARY OUTCOMES:
smoking reduction: self reported reduction | 12 months
  smoking reduction by self reported reduction

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Martín-Luján, MD, Principal Investigator — Catalan Institute of Health; Josep L Piñol-Moreso, PhD, Study Director — Catalan Institute of Health; Josep Basora-Gallisà, MD, Study Chair — Catalan Institute of Health
Locations (1):
- Jordi Gol i Gurina Foundation, Barcelona, Spain

REFERENCES:
- [Derived] Martin-Lujan F, Basora-Gallisa J, Villalobos F, Martin-Vergara N, Aparicio-Llopis E, Pascual-Palacios I, Santigosa-Ayala A, Catalin RE, Rey-Renones C, Sola R; ESPITAP Study Group Investigators. Effectiveness of a motivational intervention based on spirometry results to achieve smoking cessation in primary healthcare patients: randomised, parallel, controlled multicentre study. J Epidemiol Community Health. 2021 Oct;75(10):1001-1009. doi: 10.1136/jech-2020-216219. Epub 2021 Apr 21. PMID 33883199
- [Derived] Sorli-Aguilar M, Martin-Lujan F, Flores-Mateo G, Jardi-Pinana C, Aparicio-Llopis E, Basora-Gallisa J, Sola-Alberich R; ESPITAP Study Group investigators. Adiposity markers and lung function in smokers: a cross-sectional study in a Mediterranean population. BMC Pulm Med. 2016 Dec 9;16(1):178. doi: 10.1186/s12890-016-0341-y. PMID 27938399
- [Derived] Martin-Lujan F, Pinol-Moreso JL, Martin-Vergara N, Basora-Gallisa J, Pascual-Palacios I, Sagarra-Alamo R, Llopis EA, Basora-Gallisa MT, Pedret-Llaberia R; ESPITAP Study Group investigators. Effectiveness of a structured motivational intervention including smoking cessation advice and spirometry information in the primary care setting: the ESPITAP study. BMC Public Health. 2011 Nov 11;11:859. doi: 10.1186/1471-2458-11-859. PMID 22078490